CLINICAL TRIAL: NCT07280260
Title: Effects of Early Loading Protocol on the Survival of the Nobel N1 Implant System: A Pilot Randomized Controlled Trial
Brief Title: Clinical Performance of Nobel N1 System
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Envista (Nobel Biocare) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8328
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Tooth Loss; Dental Implant
Keywords: Tooth loss; Edentulous; Dental implants
MeSH Terms: conditions — Tooth Loss; Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: The study is a two-arm, randomized prospective clinical trial. The randomization of the patients will be done after implant has been placed and if sufficient torque was obtained as outlined previously. At this point, using a computer generated table of random numbers, patients will be randomized into early loading and delayed loading group. Since it is not possible to predict ahead of time what the final torque will be at implant placement, a third group will comprise patients that receive implants that have lower torque that cannot be randomized. These patients will follow traditional one stage or two stage protocol for implant placement and delayed protocol. Irrespective of randomization and torque status and implant placement, all patients will be followed up as part of the study and analyzed based on the group to which they belong.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early loading (Active Comparator): Delivery of the final crowns 6 weeks after the implant placement.
  Interventions: Device: Nobel N1 implant
- Delayed loading (Other): Delivery of the final crowns 12 weeks after the implant placement.
  Interventions: Device: Nobel N1 implant

INTERVENTIONS:
Device: Nobel N1 implant — A Nobel N1 implant will be placed and restored with a On 1 base

SUMMARY:
The purpose of the study is to evaluate whether N1 dental implants are successful when a final crown is placed on them at 6 weeks from implant placement surgery.

DETAILED DESCRIPTION:
This study aims to evaluate the survival and stability of the Nobel N1 dental implant and its accompanying crown over a one-year period when the crown is placed either 6 or 12 weeks after implant placement. The Nobel N1 implant is an FDA-approved, newly designed implant featuring an innovative surgical placement protocol intended to minimize bone trauma, promote faster integration, and potentially allow for the placement of final crowns earlier-at 6 weeks instead of the traditional 4 to 5 months. This study will enroll adult participants who are missing a single tooth in the back of the mouth.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 or older

  * Can provide an Informed Consent in English.
  * Absence of a single posterior tooth in mandible or maxilla with presence of natural neighboring teeth (except for second molar which only requires presence of first molar)
  * Presence of antagonist teeth
  * Possibility and will for an immediate restoration.
  * Systemic health recorded as an American Society of Anesthesiologists (ASA) I or II

Exclusion Criteria:

* · Unavailability to attend the follow-up visits.

  * A systemic contraindication for oral surgical procedures; ASA III or IV.
  * Pregnancy or nursing on screening or before the surgical procedure.
  * Diseases that could alter healing or bone metabolism (uncontrolled diabetes, diagnostic osteoporosis, etc.),
  * Taking medications that are altering healing or bone metabolism (bisphosphonates, long-time corticosteroids intake, RANK inhibitors, etc.)
  * Alcohol or drug abuse.
  * Current heavy smoking behavior (≥10 cigarettes/day).
  * Radiation therapy to the head or neck region.
  * Pathology in the implant planned sites that prevent implant placement.
  * Current diagnosis of Diabetes, which is uncontrolled (>7 HbA1C).
  * Need for sinus lift or vertical bone augmentation
  * Previously failed implant site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 6 months, 1 year
  Implant survival will be measured if it is not failed and still present at time points
Misch implant success criteria | 6 months, 1 year
  Implant success will be measured according to Misch et al.

SECONDARY OUTCOMES:
Marginal bone loss | 6 months, 1 year
  Marginal bone loss from the platform of the implant will be measured on Peri-apical X-rays and bitewings
Probing depth | 6 months, 1 year
  Probing depths will be measured at 6 surfaces
Presence of sulcular suppuration on gentle probing | 6 months, 1 year
  Presence or absence of suppuration will be evaluated upon gentle probing at 6 surfaces around the implant
Presence of sulcular bleeding on gentle probing | 6 months, 1 year
  Presence or absence of bleeding will be evaluated upon gentle probing at 6 surfaces around the implant
Peri-implant Mucosal Tissue Index | Prosthetic delivery, 6 months, 1 year
Patient satisfaction questionnaire | Prosthetic delivery, 6 months, 1 year
Prosthetic complications | 6 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- LSU School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No